CLINICAL TRIAL: NCT06954415
Title: The Clinical Application of Electrical Impedance Tomography in Clinically Ill Patients: a Cross-sectional Study
Brief Title: The Clinical Application of EIT in Clinically Ill Patients: a Cross-sectional Study
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2025-079R
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Electrical Impedance Tomography (EIT)
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention (observational study) — Questionnaire without intervention

SUMMARY:
The application of electrical impedance tomography (EIT) in intensive care is increasing. It can provide additional information on individual respiratory physiology of patients, enabling clinicians or respiratory therapists to monitor patients' respiratory responses to different ventilator settings, respiratory treatment methods or clinical evolution, and thus achieve more personalized mechanical ventilation methods. Although this technology provides a large amount of valuable information, there is still uncertainty about how to use it and interpret the results in critically ill patients. Therefore, the evidence that EIT-guided ventilation strategies can improve prognosis is still in its infancy. Through this survey, the investigators aim to understand the current experiences and guiding roles of EIT in clinical practice. The secondary objective is to learn about the current challenges of EIT in clinical and practical settings, as well as the factors that promote or hinder the implementation of EIT monitoring technology.

ELIGIBILITY:
Inclusion Criteria:

* occupation is "respiratory therapist or part-time respiratory therapy doctor/nurse";
* work city or area belongs to China;
* to complete electronic questionnaires to fill out and submit.

Exclusion Criteria:

* work city or area not belongs to China;
* The questionnaire is not completed or quit midway;
* Other invalid questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Doctors/respiratory therapists with experience in EIT application in Chinese intensive care units
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of EIT usage | Baseline